CLINICAL TRIAL: NCT03618966
Title: Neuromuscular Magnetic Stimulation Counteracts Muscle Decline in ALS Patients
Brief Title: Neuromuscular Magnetic Stimulation in ALS Patients
Acronym: NMS-ALS
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Roma La Sapienza (Other)
Responsible Party: Principal Investigator, Maurizio Inghilleri, Associate Professor, University of Roma La Sapienza
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 2174
Record Dates: First submitted 2018-07-23; First posted 2018-08-07 (Actual); Last update posted 2018-08-07 (Actual); Status verified 2018-08

CONDITIONS: Amyotrophic Lateral Sclerosis
Keywords: Amyotrophic lateral sclerosis; Muscle disease; Neuromuscular magnetic stimulation
MeSH Terms: conditions — Amyotrophic Lateral Sclerosis; Muscular Diseases

STUDY DESIGN:
Intervention Model Description: Patients will be randomized in two groups by receiving a sequential number according to a from a computer-generated random list. A first group will receive a real stimulation (rNMMS) of the right arm and a sham stimulation (sNMMS) of the left arm; a second group received a rNMMS of the left arm and a sNMMS of the right arm. Every cycle of stimulation will last two weeks. All patients will undergo a medial nerve conduction study (NCS) and a clinical evaluation before and at the end of the treatment and another evaluation after two weeks after the end of treatment. Clinical examination will include i) handgrip strength test for the measure of maximal isometric strength of hand and flexor forearm muscles; ii) MRC Muscle Scale for manual muscular testing of the upper limbs. At the end of the stimulation procedure, a needle muscle biopsy under a local anesthetic will be performed bilaterally from flexor carpi radialis muscle for histological, physiological and molecular studies.
Who Masked: Participant, Care Provider, Investigator
Masking Description: All the electrophysiological experiments will be performed in double-blind fashion.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Right-real NMMS Group (Experimental): It will receive a real stimulation (rNMMS) of the right arm and a sham stimulation (sNMMS) of the left arm
  Interventions: Device: Neuromuscular magnetic stimulation (NMMS)
- Left-real NMMS Group (Active Comparator): It will receive a rNMMS of the left arm and a sNMMS of the right arm
  Interventions: Device: Neuromuscular magnetic stimulation (NMMS)

INTERVENTIONS:
Device: Neuromuscular magnetic stimulation (NMMS) — It is a non-invasive, stimulation technique that does not induce high-intensity cutaneous electric fields and does not activate skin nociceptors, thus resulting in a painless and better-tolerated procedure. rNMMS is delivered through a high-frequency magnetic stimulator connected to a conventional circular cooled coil. Magnetic stimulator is placed above the flexor muscles of the forearm. rNMMS is delivered at a 5-Hz frequency and with a 100% stimulation intensity of 100% of the maximum intensity in 140 trains of 50 stimuli. sNMMS is delivered with a sham coil producing similar acoustic sensations and mechanical skin perceptions.

SUMMARY:
Aim of the study is to verify whether neuromuscular magnetic stimulation can improve muscle function in spinal-onset Amyotrophic Lateral Sclerosis (ALS) patients.

DETAILED DESCRIPTION:
Background: Amyotrophic lateral sclerosis (ALS) is a multi-factorial and multi-systemic pathology associated with motor neuron degeneration, muscle atrophy and paralysis. Mounting evidence suggests that the earliest presymptomatic functional and pathological changes are occurring distally in axons and at the neuromuscular junction (NMJ). These changes precede, and can be independent of the loss of cell bodies or alterations in other cell types already linked to the ALS disease process. In line with these studies, we found that in human ALS muscles the acetylcholine receptors (AChRs) are less sensitive to ACh than denervated non-ALS muscles. It has been also reported that muscle specific expression of mutant superoxide dismutase (SOD1) gene induces muscle atrophy, significant reduction in muscle strength, mitochondrial dysfunction, microgliosis, and neuronal degeneration, suggesting that retrograde signals from muscle to nerve may contribute to synapse and axon damage. This suggests that skeletal muscle is an important target for therapeutic intervention. Neuromuscular system may be artificially stimulated either by an electrical stimulation (ES) or by time-varying electromagnetic fields. Neuromuscular magnetic stimulation (NMMS) has been proposed as an alternative, non-invasive, stimulation technique.

Objective: aim of the study is to verify whether neuromuscular magnetic stimulation can improve muscle function in spinal-onset Amyotrophic Lateral Sclerosis (ALS) patients. We will study if neuromuscular magnetic stimulation can counteract muscle atrophy by promoting the modulation of factors associated with muscle catabolism and/or increasing the efficacy of nicotinic acetylcholine receptors.

Methods: At the baseline visit, ALS patients will be randomized in two groups to receive daily real neuromuscular magnetic stimulation in one arm and sham neuromuscular magnetic stimulation in the opposite arm for two weeks. All patients will undergo median nerve conduction study and a clinical examination, including handgrip strength test and evaluation of upper limbs muscle strength by Medical Research Council Muscle Scale. At the end of the stimulation procedures, a needle muscle biopsy will be performed bilaterally from flexor carpi radialis muscle. Muscle samples will be used to perform histomorphometric and molecular analysis and electrophysiological recordings of acetylcholine evoked currents.

ELIGIBILITY:
Inclusion Criteria:

* diagnosis of probable or definite ALS with spinal-onset
* right-handed patients
* a bilateral symmetric muscular deficit in flexor carpi radialis muscle or flexor digitorum profundus muscle (defined by a MRC Muscle Scale score of 3-4/5)

Exclusion Criteria:

* history of epilepsy or severe headaches,
* pregnancy or breast-feeding
* patients with implanted cardiac pacemaker, neurostimulators, surgical clips or medical pumps
* presenting any other comorbid condition affecting the possibility of completing the study

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2014-11-01 (Actual); Primary Completion 2016-05-01 (Actual); Study Completion 2017-11-01 (Actual)

PRIMARY OUTCOMES:
Change from baseline to Week 2 in the muscle strength measured by Medical Research Council Muscle Scale (MRC). | Baseline to Week 2
  Evaluation of the efficacy of NMMS in improving the muscular strength in ALS patients as measured by MRC-score (numeric scale, normal value: 35 for upper limbs, 40 for lower limbs).

SECONDARY OUTCOMES:
Change from baseline to Week 2 in the muscle strength measured by handgrip dynamometry | Baseline to Week 2
  Evaluation of the efficacy of NMMS in improving the muscular strength in ALS patients as measured by handgrip dynamometry (numeric scale, normal value: >35 for female, >45 for male)
Change from baseline to Week 2 in the Compound Muscle Action Potential (CMAP) amplitude from flexor carpi radialis | Baseline to Week 2
  Evaluation of the effect of NMMS on the electrophysiological parameter (CMAP) to analyse the physiological mechanisms of the applied neurophysiological technique (milliVolt, mV, normal value 10.2 mV).
Change from baseline to Week 2 in the amplitude of the ACh-evoked currents (IACh) for nicotinic acetylcholine receptors | Baseline to Week 2
  Evaluation of the effect of NMMS on the nicotinic acetylcholine receptor in patients with ALS (nanoAmpere, nA)
Change from baseline to Week 2 on levels of insulin-like growth factor-1 (IGF-1) and Myostatin | Baseline to Week 2
  Evaluation of the effect of NMMS on the adaptation changes of gene expression due to rNMMS quantifying shifts in messenger ribonucleic acid (mRNA) levels of a selected panel of genes involved in muscle growth (numeric value)
Change from baseline to Week 2 on the diameter size of muscle fibers | Baseline to Week 2
  Evaluation of the effect of NMMS on histomorphometric analysis in ALS muscle fibers (micrometer, μm).
Change from baseline to Week 2 on levels of Muscle Atrophy F-box (MAFbx)/Atrogin-1 and Muscle Ring-Finger Protein 1 (MuRF-1) | Baseline to Week 2
  Evaluation of the effect of NMMS on the adaptation changes of gene expression due to rNMMS quantifying shifts in mRNA levels of a selected panel of genes involved in downregulation of atrophy-related genes (numeric value)

CONTACTS AND LOCATIONS:
Overall Officials: Maurizio Inghilleri, Prof, Principal Investigator — Department of Human Neuroscience, Umberto I Hospital-University of Rome Sapienza

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Musaro A. Understanding ALS: new therapeutic approaches. FEBS J. 2013 Sep;280(17):4315-22. doi: 10.1111/febs.12087. Epub 2013 Jan 3. PMID 23217177
- [Background] Taylor JP, Brown RH Jr, Cleveland DW. Decoding ALS: from genes to mechanism. Nature. 2016 Nov 10;539(7628):197-206. doi: 10.1038/nature20413. PMID 27830784
- [Background] Dadon-Nachum M, Melamed E, Offen D. The "dying-back" phenomenon of motor neurons in ALS. J Mol Neurosci. 2011 Mar;43(3):470-7. doi: 10.1007/s12031-010-9467-1. Epub 2010 Nov 7. PMID 21057983
- [Background] Dupuis L, Loeffler JP. Neuromuscular junction destruction during amyotrophic lateral sclerosis: insights from transgenic models. Curr Opin Pharmacol. 2009 Jun;9(3):341-6. doi: 10.1016/j.coph.2009.03.007. Epub 2009 Apr 20. PMID 19386549
- [Background] Dobrowolny G, Aucello M, Rizzuto E, Beccafico S, Mammucari C, Boncompagni S, Belia S, Wannenes F, Nicoletti C, Del Prete Z, Rosenthal N, Molinaro M, Protasi F, Fano G, Sandri M, Musaro A. Skeletal muscle is a primary target of SOD1G93A-mediated toxicity. Cell Metab. 2008 Nov;8(5):425-36. doi: 10.1016/j.cmet.2008.09.002. PMID 19046573
- [Background] Loeffler JP, Picchiarelli G, Dupuis L, Gonzalez De Aguilar JL. The Role of Skeletal Muscle in Amyotrophic Lateral Sclerosis. Brain Pathol. 2016 Mar;26(2):227-36. doi: 10.1111/bpa.12350. PMID 26780251
- [Background] Palma E, Inghilleri M, Conti L, Deflorio C, Frasca V, Manteca A, Pichiorri F, Roseti C, Torchia G, Limatola C, Grassi F, Miledi R. Physiological characterization of human muscle acetylcholine receptors from ALS patients. Proc Natl Acad Sci U S A. 2011 Dec 13;108(50):20184-8. doi: 10.1073/pnas.1117975108. Epub 2011 Nov 29. PMID 22128328
- [Background] Palma E, Reyes-Ruiz JM, Lopergolo D, Roseti C, Bertollini C, Ruffolo G, Cifelli P, Onesti E, Limatola C, Miledi R, Inghilleri M. Acetylcholine receptors from human muscle as pharmacological targets for ALS therapy. Proc Natl Acad Sci U S A. 2016 Mar 15;113(11):3060-5. doi: 10.1073/pnas.1600251113. Epub 2016 Feb 29. PMID 26929355
- [Background] Kern H, Barberi L, Lofler S, Sbardella S, Burggraf S, Fruhmann H, Carraro U, Mosole S, Sarabon N, Vogelauer M, Mayr W, Krenn M, Cvecka J, Romanello V, Pietrangelo L, Protasi F, Sandri M, Zampieri S, Musaro A. Electrical stimulation counteracts muscle decline in seniors. Front Aging Neurosci. 2014 Jul 24;6:189. doi: 10.3389/fnagi.2014.00189. eCollection 2014. PMID 25104935
- [Background] Eusebi F, Palma E, Amici M, Miledi R. Microtransplantation of ligand-gated receptor-channels from fresh or frozen nervous tissue into Xenopus oocytes: a potent tool for expanding functional information. Prog Neurobiol. 2009 May;88(1):32-40. doi: 10.1016/j.pneurobio.2009.01.008. Epub 2009 Feb 7. PMID 19428960
- [Background] Musaro A, McCullagh K, Paul A, Houghton L, Dobrowolny G, Molinaro M, Barton ER, Sweeney HL, Rosenthal N. Localized Igf-1 transgene expression sustains hypertrophy and regeneration in senescent skeletal muscle. Nat Genet. 2001 Feb;27(2):195-200. doi: 10.1038/84839. PMID 11175789
- [Background] Scicchitano BM, Rizzuto E, Musaro A. Counteracting muscle wasting in aging and neuromuscular diseases: the critical role of IGF-1. Aging (Albany NY). 2009 May 13;1(5):451-7. doi: 10.18632/aging.100050. PMID 20157530
- [Background] Trendelenburg AU, Meyer A, Rohner D, Boyle J, Hatakeyama S, Glass DJ. Myostatin reduces Akt/TORC1/p70S6K signaling, inhibiting myoblast differentiation and myotube size. Am J Physiol Cell Physiol. 2009 Jun;296(6):C1258-70. doi: 10.1152/ajpcell.00105.2009. Epub 2009 Apr 8. PMID 19357233